CLINICAL TRIAL: NCT05506358
Title: Evaluation of Low-cost Techniques for Detecting Sickle Cell Disease and β-thalassemia in Nepal and Canada
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Boris Stoeber, Professor in the Department of Electrical and Computer Engineering and in the Department of Mechanical Engineering, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H22-00294; 85/2022 (Other: Nepal Health Research Council); H22-00294 (Other: UBC Clinical Research Ethics Board); H21-01929 (Other: UBC-Providence Health Care Research Institute)
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Sickle Cell Disease; Sickle Cell Trait; Beta-Thalassemia; Sickle Cell-Beta Thalassemia; Sickle Cell-SS Disease
Keywords: low-cost test; point-of-care diagnostics; automated sickling test; solubility test; HemoTypeSC; Sickle Scan; Gazelle Hb Variant Test; Machine learning; Image database; Red blood cells
MeSH Terms: conditions — Anemia, Sickle Cell; Sickle Cell Trait; beta-Thalassemia

STUDY DESIGN:
Intervention Model Description: Around 90 participants will be recruited in Canada - 30 with SCD (HbSS), 30 with SCT (HbAS), and 30 healthy participants (HbAA).
  Around 120 participants will be recruited in Nepal - 20 with SCD (HbSS), 20 with SCT (HbAS), 20 with sickle cell / β-thalassaemia compound heterozygous form (HbS/β-thalassemia), 20 with β-thalassaemia (Hbβ/ β-thalassemia), 20 with β-thalassaemia trait or carrier form (HbA/β-thalassemia), and 20 healthy participants (HbAA).
  3-4 mL of blood will be drawn using standard phlebotomy practices. The following tests will be performed:
  a. Low-cost tests i. Sickling test with low-cost microscope and automated screening with machine learning ii. Sickling test with traditional microscope (conventional manual screening used in Nepal) iii. HbS solubility test iv. Commercial point-of-care assays (HemoTypeSC and Sickle SCAN) v. Gazelle Hb variant test
  b. Gold standard test: HPLC, for determining the accuracies of low-cost screening techniques
Masking Description: All the participants and study team members will be informed of the tests and devices used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 1) HbSS; 2) HbAS; 3) HbS/β-thalassemia; 4)Hbβ/β-thalassemia; 5) HbA/β- thalassemia; 6) HbAA (Other): Around 20 participants each (in Nepal):
  * with the homozygous form of sickle cell disease (HbSS)
  * with the heterozygous form of sickle cell disease (HbAS)
  * with the compound heterozygous form of sickle cell disease (HbS/β-thalassemia)
  * with the carrier form of β-thalassemia (HbA/β-thalassemia)
  * with the carrier form of β-thalassemia (HbA/β-thalassemia)
  * without any known hemoglobin disorders, such as sickle cell disease, sickle cell trait, β-thalassemia, etc.
  Around 30 participants each (in Canada):
  * with the homozygous form of sickle cell disease (HbSS)
  * with the heterozygous form of sickle cell disease (HbAS)
  * without any known hemoglobin disorders, such as sickle cell disease, sickle cell trait, β-thalassemia, etc.
  Interventions: Diagnostic Test: High performance liquid chromatography; Device: Automated sickling test; Diagnostic Test: HbS solubility test; Device: HemoTypeSC; Device: Sickle SCAN; Device: Gazelle Hb Variant Test

INTERVENTIONS:
Diagnostic Test: High performance liquid chromatography — High performance liquid chromatography (HPLC) using the D10 System by Bio-Rad Laboratories will be used as the gold standard test.
Device: Automated sickling test — The standard sickling test using 2% sodium metabisulphite will be augmented using an automated microscope (such as Octopi) and machine learning, and will be used as one of the low-cost tests.
Diagnostic Test: HbS solubility test — Standard HbS solubility test currently used in Nepal (e.g. Sicklevue) will be used as one of the low-cost tests
Device: HemoTypeSC — A point-of-care lateral flow assay, HemoTypeSC (https://www.hemotype.com/), will be used as one of the low-cost tests
Device: Sickle SCAN — A point-of-care lateral flow assay, Sickle SCAN (https://www.biomedomics.com/products/hematology/sicklescan/), will be used as one of the low-cost tests
Device: Gazelle Hb Variant Test — A portable electrophoresis machine, Gazelle diagnostic device (https://hemexhealth.com/), will be used as one of the low-cost tests

SUMMARY:
Sickle cell disease (SCD) is an inherited blood disorder associated with acute illness and organ damage. In high resource settings, early screening and treatment greatly improve quality of life. In low resource settings, however, mortality rate for children is high (50-90%). Low-cost and accurate screening techniques are critical to reducing the burden of the disease, especially in remote/rural settings. The most common and severe form of SCD is sickle cell anemia (SCA), caused by the inheritance of genes causing abnormal forms of hemoglobin (called sickle hemoglobin or hemoglobin S) from both parents. The asymptomatic or carrier form of the disease, known as sickle cell trait (SCT), is caused by the inheritance of only one variant gene from one of the parents. In areas such as Nepal, β-thalassemia (another inherited blood disorder) and SCD are both prevalent, and some combinations of these diseases lead to severe symptoms.

The purpose of this study is to determine the accuracy of low-cost point-of-care techniques for screening and detecting sickle cell disease, sickle cell trait, and β-thalassaemia, which will subsequently inform on feasible solutions for detecting the disease in rural, remote, or low-resource settings. One of the goals of the study is to evaluate the feasibility of techniques, such as the sickling test with low-cost microscopy and machine learning, HbS solubility test, commercial lateral-flow assays (HemoTypeSC and Sickle SCAN), and the Gazelle Hb variant test, to supplement or replace gold standard tests (HPLC or electrophoresis), which are expensive, require highly trained personnel, and are not easily accessible in remote/rural settings.

The investigators hypothesize that:

1. an automated sickling test (standard sickling test enhanced using low-cost microscopy and machine learning) has a higher overall accuracy than conventional screening techniques (solubility and sickling tests) to detect hemoglobin S in blood samples
2. the automated sickling test can additionally classify SCD, SCT and healthy individuals with a sensitivity greater than 90%, based on morphology changes of red blood cells, unlike conventional sickling or solubility tests that do not distinguish between SCD and SCT cases
3. Gazelle diagnostic device can detect β-thalassaemia and SCD/SCT with an overall accuracy greater than 90%, compared with HPLC as the reference test

DETAILED DESCRIPTION:
Overall, the hypothesis is that an assessment of the performance and accuracies of low-cost point-of-care techniques (automated sickling test, solubility test, lateral-flow assays, Gazelle Hb variant test) against HPLC tests will provide researchers and health workers with feasible alternative options for screening and detecting SCD, SCT and β-thalassaemia in a variety of situations based on the needs of the communities and the resources available.

Objectives

Objectives specific to the current study are to:

1. Determine accuracy (sensitivity and specificity) of automated sickling test to detect HbS, compared to gold standard HPLC, and to conventional solubility test
2. Determine whether SCD, SCT and healthy individuals can be classified using the automated sickling test that leverages machine learning on images of blood films under hypoxia
3. Validate accuracy (>95% sensitivity and specificity) of lateral- flow assays (HemoTypeSC and Sickle SCAN) to detect SCD/SCT, and of Gazelle variant test to detect SCD, SCT, and β-thalassaemia; and determine if low-cost techniques can potentially replace HPLC/electrophoresis tests in rural and remote settings

Long-term objectives of the overall project are to:

1. Implement trained machine learning algorithm to classify SCD, SCT and healthy individuals during screening tests in Nepal
2. Implement relevant low-cost point-of-care techniques in rural and remote communities of Nepal using insights and conclusions from current study

The plan of the study to screen the communities (e.g. in Nepalgunj, in Vancouver) using the following:

a. Low-cost screening i. Sickling test with low-cost microscope and automated screening with machine learning ii. Sickling test with traditional microscope (conventional manual screening used in Nepal) iii. HbS solubility test iv. Commercial point-of-care assays (HemoTypeSC and Sickle SCAN) v. Gazelle Hb variant test b. Gold standard test: HPLC, for determining the accuracies of low-cost screening techniques

De-identified data (images of blood films and associated documentation) will also be deposited in an online public repository, such as the Federated Research Data Repository (FRDR). FRDR is a service of the Digital Research Alliance of Canada (Alliance), a not-for-profit organization that supports digital research infrastructure in Canada. FRDR is hosted on national infrastructure, managed and administered by the Digital Research Alliance of Canada.

ELIGIBILITY:
Inclusion Criteria:

Since the techniques evaluated in the study aims at detecting sickle cell disease (SCD), sickle cell trait (SCT), and β- thalassemia, the following number of participants will be included in Nepal:

* 20 individuals with SCD (HbSS)
* 20 individuals with SCT (HbAS)
* 20 individuals with sickle cell/β-thalassemia compound heterozygous form (HbS/β-thalassemia)
* 20 individuals with β-thalassemia (Hbβ/β-thalassemia)
* 20 individuals with β-thalassemia trait or carrier form (HbA/β- thalassemia)
* 20 healthy individual participants or normal participants (HbAA, participants without any known hemoglobin disorders, such as SCD, SCT or β-thalassemia)

The following number of participants will be included in Canada:

* 30 individuals with SCD (HbSS)
* 30 individuals with SCT (HbAS)
* 30 healthy individual participants or normal participants (HbAA, participants without any known hemoglobin disorders, such as SCD, SCT or β-thalassemia)

Participants older than 1 year of age at the time of drawing blood will be eligible. Signed and dated consent or assent forms will be required by the participants or their parents/guardians.

Exclusion Criteria:

The exclusion criteria for the study:

* Transfusion within the last 3 months
* Pregnancy Participants who wish to withdraw from the study will also be excluded.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Stoeber, Principal Investigator — University of British Columbia
Locations (3):
- Canada (2):
  - BC Children's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
- Mount Sagarmatha Polyclinic and Diagnostic Center, Nepalgunj, Banke, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data and test results will be shared. The test results for the low-cost tests and HPLC tests will be published in aggregate form. De-identified images of blood films will be deposited in an online public repository, such as Federated Research Data Repository (FRDR).

REFERENCES:
- [Derived] Shrestha P, Lohse H, Bhatla C, McCartney H, Alzaki A, Sandhu N, Oli PK, Chaudhary S, Amid A, Onell R, Au N, Merkeley H, Kapoor V, Pande R, Stoeber B. Evaluation of low-cost techniques to detect sickle cell disease and beta-thalassemia: an open-label, international, multicentre study. Lancet Reg Health Southeast Asia. 2025 Mar 29;35:100571. doi: 10.1016/j.lansea.2025.100571. eCollection 2025 Apr. PMID 40230447

RESULTS

PARTICIPANT FLOW:
Groups:
- HbSS: HbSS: homozygous form of sickle cell disease
- HbAS: HbAS: heterozygous (carrier) form of sickle cell disease
- HbS/β-thalassemia: HbS/β-thalassemia: compound heterozygous form of sickle cell disease (with β-thalassemia)
- HbA/β-thalassemia: HbA/β-thalassemia: β-thalassemia trait (carrier form)
- HbAA: HbAA: participants without any known hemoglobin disorders, such as sickle cell disease, sickle cell trait, β-thalassemia, etc.
Period: Overall Study
Arm/Group | HbSS | HbAS | HbS/β-thalassemia | HbA/β-thalassemia | HbAA
Started | 33 | 45 | 11 | 26 | 30
Completed | 29 | 45 | 11 | 23 | 30
Not Completed | 4 | 0 | 0 | 3 | 0
Not completed — Sickle cell disease with transfusion within 3 months | 2 | 0 | 0 | 0 | 0
Not completed — Sickle cell disease with Hereditary persistence of fetal hemoglobin (HPFH) | 2 | 0 | 0 | 0 | 0
Not completed — Beta-thalassemia major with transfusion within 2 months | 0 | 0 | 0 | 1 | 0
Not completed — Sample hemolysis observed under the microscope | 0 | 0 | 0 | 1 | 0
Not completed — HbE trait | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Note that the demographic information (age, sex) is reported for all different groups combined, and individual analysis of age and sex distribution per group is not performed due to the way the data was collected. In Canada, only averages and ranges for age and sex were collected rather than distribution per group.
Groups:
- 1) HbSS; 2) HbAS; 3) HbS/β-thalassemia; 4) HbA/β-thalassemia; 5) HbAA: Please note that the demographic information (age, sex) is reported for all different groups combined, and individual analysis of age and sex distribution per group is not performed due to the way the data was collected. In Canada, only averages and ranges for age and sex were collected rather than distribution per group.
  Number of participants considered in the study:
  29 HbSS: homozygous form of sickle cell disease 45 HbAS: heterozygous (carrier) form of sickle cell disease 11 HbS/β-thalassemia: compound heterozygous form of sickle cell disease (with β-thalassemia) 23 HbA/β-thalassemia: β-thalassemia trait (carrier form) 30 HbAA: participants without any known hemoglobin disorders, such as sickle cell disease, sickle cell trait, β-thalassemia, etc.
Arm/Group | 1) HbSS; 2) HbAS; 3) HbS/β-thalassemia; 4) HbA/β-thalassemia; 5) HbAA
Number analyzed (Participants) | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33
  Between 18 and 65 years | 103
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 27
  Nepal | 111

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity, Specificity, Positive Predictive Value and Negative Predictive Value
Description: The following metrics will be determined for the low-cost tests to be evaluated as indicated below (where TP = true positive, TN = true negative, FP = false positive, FN = false negative):
  1. Sensitivity = TP/(TP + FN)
  2. Specificity = TN/(FP + TN)
  3. Positive predictive value = TP/(TP + FP)
  4. Negative predictive value = TN/(TN + FN)
  These metrics will be calculated for the low-cost technologies against the reference test, HPLC, for detecting the presence of sickle hemoglobin and β- thalassemia. The low-cost technologies include automated sickling test (standard sickling test enhanced using low-cost microscopy and machine learning), solubility test, HemoTypeSC, Sickle SCAN, and Gazelle Hb Variant test. The test results of the low-cost technologies will be compared with those of the reference test to get the values of TP, TN, FP and FN, which will then be used to calculate the metrics listed above.
Time Frame: baseline
Measure: Number; unit: percentage
Arm/Group | HbSS | HbAS | HbS/β-thalassemia | HbA/β-thalassemia | HbAA
Number analyzed (Participants) | 29 | 45 | 11 | 23 | 30
percentage
  Gazelle (sensitivity) | 96.6 | 100 | 0 | 91.3 | 96.7
  Gazelle (specificity) | 89.9 | 100 | 99.2 | 99.1 | 98.1
  Gazelle (PPV) | 71.8 | 100 | 0 | 95.5 | 93.5
  Gazelle (NPV) | 99 | 100 | 92 | 98.3 | 99.1
  HemoTypeSC (sensitivity) | 100 | 97.8 | 0 | 0 | 100
  HemoTypeSC (specificity) | 89 | 100 | 100 | 100 | 78.7
  HemoTypeSC (NPV) | 100 | 98.9 | 92 | 83.3 | 100
  Sickle SCAN (sensitivity) | 100 | 100 | 0 | 0 | 100
  Sickle SCAN (specificity) | 89.9 | 100 | 100 | 100 | 78.7
  Sickle SCAN (NPV) | 100 | 100 | 92 | 83.3 | 100

ADVERSE EVENTS:
Time Frame: 1 day
Description: Blood collection for all participants followed normal phlebotomy practices in the clinic and hospital. The participants were observed for potential risks of phlebotomy such as:
  1. Excessive bleeding
  2. Fainting or lightheadedness
  3. Hematoma or blood accumulating under the skin
  4. Infection from blood borne pathogens
  5. Multiple punctures to locate veins
Arm/Group | HbSS | HbAS | HbS/β-thalassemia | HbA/β-thalassemia | HbAA
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/45 | 0/11 | 0/23 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/45 | 0/11 | 0/23 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/45 | 0/11 | 0/23 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT05506358/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT05506358/ICF_001.pdf